CLINICAL TRIAL: NCT06004401
Title: The Observation on the Efficacy of Dual Therapy Based on Vonoprazan in Eradicating Helicobacter Pylori
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Wei-Fen Xie, Head of gastroenterology，Shanghai Changzheng Hospital, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CZHX2023.07
Record Dates: First submitted 2023-07-30; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: The Eradication Rate of Helicobacter Pylori

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Penicillin negative test group (Experimental): （Vonopazan 20mg 2//day+Amoxicillin 1.0g 3/day）*14 days
  Interventions: Drug: Vonopazan +Amoxicillin
- Penicillin negative contral group (Active Comparator): （Rabeprazole tablets 10mg 2/day+colloidal pectin bismuth 200mg 2/day+Amoxicillin 1g 2/day+Clarithromycin 500mg 2/day）*14 days
  Interventions: Drug: Rabeprazole +colloidal pectin bismuth +Amoxicillin +Clarithromycin
- Penicillin positive test group (Experimental): （Vonopazan 20mg 2/day+Minocycline 100mg 2/day）*14 days
  Interventions: Drug: Vonopazan +Minocycline
- Penicillin positive control group (Active Comparator): （Rabeprazole tablets 10mg 2/day+colloidal pectin bismuth 200mg 2/day+Metronidazole 0.4g 3/day+Clarithromycin 500mg 2/day）*14 days
  Interventions: Drug: Rabeprazole +colloidal pectin bismuth +Metronidazole +Clarithromycin

INTERVENTIONS:
Drug: Vonopazan +Amoxicillin — Vonopazan 20mg 2//day+Amoxicillin
  Arms: Penicillin negative test group
Drug: Rabeprazole +colloidal pectin bismuth +Amoxicillin +Clarithromycin — Rabeprazole tablets 10mg 2/day+colloidal pectin bismuth 200mg 2/day+Amoxicillin 1g 2/day+Clarithromycin 500mg 2/day
  Arms: Penicillin negative contral group
Drug: Vonopazan +Minocycline — Vonopazan 20mg 2/day+Minocycline 100mg 2/day
  Arms: Penicillin positive test group
Drug: Rabeprazole +colloidal pectin bismuth +Metronidazole +Clarithromycin — Rabeprazole tablets 10mg 2/day+colloidal pectin bismuth 200mg 2/day+Metronidazole 0.4g 3/day+Clarithromycin 500mg 2/day
  Arms: Penicillin positive control group

SUMMARY:
Helicobacter pylori（Hp）is listed as a Class 1 carcinogen by the International Agency for Research of Cancer (IARC), Eradicating Hp can significantly reduce the risk of gastric cancer. In recent years, the resistance rate of Hp to antibiotics, especially Clarithromycin and Metronidazole, has increased, leading to the gradual reduction of the eradication rate . In addition, PPI is mainly metabolized by CYP2C19 in the body, and the genetic polymorphism of this enzyme activity in the population results in significant individual differences in the acid suppression effect of PPI; At the same time, PPI will affect the metabolism of other drugs by affecting the activity of CYP2C19 in the liver.

Potassium ion competitive acid blockers (P-CABs) are a new type of antacids, and vonoprazan is a representative of this class of drugs. Compared to traditional proton pump inhibitors, it has higher selectivity towards proton pumps, stronger acid inhibition effect, faster onset time , longer sustained acid inhibition time, and less influence from food consumption. Therefore, it can effectively eliminate Helicobacter pylori . In recent years, Vonoprazan has been widely used in the eradication treatment of Hp . Vonoprazan can inhibit gastric acid secretion more strongly and persistently, therefore, eradication plans based on vonoprazan are expected to improve the eradication rate of Hp.

Related studies have shown that compared to traditional proton pump inhibitors, vonoprazan has a more significant therapeutic effect and higher safety in the treatment of Helicobacter pylori positive peptic ulcers due to its unique mechanism of action..In recent years, there have been reports of successful eradication of multi drug resistant Hp retreated patients with Semisynthesis tetracycline. Some domestic scholars are also gradually trying to use Semisynthesis tetracycline to eradicate Hp infection. Minocycline is a Semisynthesis tetracycline. The drug sensitivity test in vitro showed that the resistance rate of Hp to Minocycline was low , suggesting that Minocycline may have a better effect on eradicating Hp.

Therefore, the investigators further carried out a prospective single center clinical study and set up a penicillin negative group. One month after treatment, 13C carbon breath test was performed to check the efficacy, in order to explore the efficacy of the combination therapy based on vonoprazan in eradicating Hp, especially whether it is a good choice for penicillin allergy.

DETAILED DESCRIPTION:
After one month of treatment, a 13C carbon breath test was conducted to investigate the efficacy of a dual therapy based on vorolaxen in eradicating Hp, especially for those allergic to penicillin.

ELIGIBILITY:
Inclusion Criteria:•

1. Male or female aged 18-75;
2. Initial treatment patients with Helicobacter pylori infection (positive 13C carbon breath test/positive Hp in gastroscopy pathological biopsy);
3. Not taking antibiotics, bismuth agents, or traditional Chinese medicine with antibacterial effects (Isatis indigotica, berberine, honeysuckle, forsythia suspensa) in the first 4 weeks; I did not take drugs that affect Hp activity such as PPI or H2 receptor antagonists in the first two weeks.

   -

   Exclusion Criteria:
   * 1）Age<18 years old or>75 years old; 2）Pregnant and lactating women; 3）Patients with severe primary diseases such as cardiovascular, liver, kidney, and hematopoietic systems, as well as mental illness.

     4）History of Drug allergy used in the treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-08-20 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The eradication rate of Helicobacter pylori | two years
  whether the dual therapy based on vorolaxen has advantages over traditional quadruple therapy in penicillin negative and positive patients

IPD SHARING:
Plan to Share IPD: No